CLINICAL TRIAL: NCT01118572
Title: A Phase III Study of YM177 (Postoperative Pain) -- An Etodolac- and Placebo-controlled, Multicenter, Double-blind, Group Comparison Study to Verify the Efficacy of YM177 (Celecoxib) in Postoperative Pain Patients --
Brief Title: A Study to Verify the Efficacy of YM177 (Celecoxib) in Postoperative Pain Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 177-CL-102
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Post Operative Pain
Keywords: Celecoxib; Celecox; Pain; Surgery; NSAIDs
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Celecoxib; Etodolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- YM177 group (Experimental)
  Interventions: Drug: YM177
- etodolac group (Active Comparator)
  Interventions: Drug: etodolac
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YM177 — oral
  Other Names: Celecoxib; Celecox
  Arms: YM177 group
Drug: etodolac — oral
  Other Names: Osteluc; Hypen
  Arms: etodolac group
Drug: Placebo — oral
  Arms: placebo group

SUMMARY:
Aim of the study is to compare efficacy and safety of YM177 with placebo and etodolac in patients with postoperative pain.

DETAILED DESCRIPTION:
To verify the superiority to placebo and the noninferiority to etodolac of YM177 in terms of efficacy assessment in patients with postoperative pain. Also, to compare them in terms of safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous pain within 24 hours postoperatively
* The intensity of the pain:

  * 4-categorical assessment: "Moderate pain" or "Severe pain"
  * VAS assessment: 45.0 mm or higher
* Patients whose postoperative pain can be managed using an oral NSAID

Exclusion Criteria:

* A past history of aspirin-induced asthma
* A past of ischemic heart disease, serious arrhythmia, congestive heart failure or cerebrovascular disease
* Patients who undergoes the surgical procedure under general anesthesia
* Patients taking excluded medications

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Patient impressions (4-categorical assessments) | For 2 days

SECONDARY OUTCOMES:
Pain intensity | For 2 days
Pain intensity difference | For 2 days
Discontinuation due to insufficient efficacy | For 2 days
Safety assessed by AE, clinical lab tests and vital signs | For 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyusyu
  - Shikoku
  - Tōhoku